CLINICAL TRIAL: NCT01569646
Title: Significance of Monocytosis and Culprit Vessel in Patients With Acute ST Elevation Myocardial Infarction
Brief Title: Monocytosis and Culprit Vessel in STEMI Patients
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 08-021
Record Dates: First submitted 2010-06-02; First posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: STEMI
Keywords: monocytes; culprit vessels
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Increased white blood cell count at the onset of an acute ST elevation myocardial infarction has been shown to be associated of increased incidence of heart failure and mortality. Now monocytes which are a subset of white blood cells may have a prognostic value for patients presenting with acute ST segment elevation myocardial infarction. A monocyte count of greater than 800/mm3 following acute myocardial infarction has been shown to be associated with increased incidence of left ventricular dysfunction. The investigators study would retrospectively collect data on patients with ST elevation myocardial infarction, looking for an association between high monocyte count and the culprit vessel causing the myocardial infarction. The investigators would also investigate whether monocytosis would be a marker of poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* STEMI

Exclusion Criteria:

* Patients on antibiotics and steroids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: STEMI patients,
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2008-04

PRIMARY OUTCOMES:
Association between monocyte count and culprit vessel | 1 day

SECONDARY OUTCOMES:
clinical outcomes of troponin and monocyte in stemi patients | 0 - 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Duccio Baldari, MD, FACC, Principal Investigator — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States